CLINICAL TRIAL: NCT06765954
Title: Open-Label, Phase 2 Clinical Trial of Pre-Radiation and Post-Radiation Immunotherapy With N-803, ETBX-071, and M-CENK in Combination With Radiation for Participants With High-Risk Prostate Cancer
Brief Title: Immunotherapy With N 803, ETBX-071, and M-CENK in Combination With Radiation for Participants With High-Risk Prostate Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ResQ110B-PROS
Record Dates: First submitted 2024-12-20; First posted 2025-01-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-12

CONDITIONS: High-risk Prostate Cancer
Keywords: high-risk prostate cancer; Prostate Cancer; N-803; ETBX-071; M-CENK; Radiation Therapy/EBRT; Combination Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ALT-803; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: While the treatment involves multiple stages (pre-radiation immunotherapy, radiation, post-radiation immunotherapy), participants are assigned to one arm of the study and receive the complete treatment regimen within that arm. There's no crossover or other complex design element described; participants receive a consistent set of interventions according to their assigned group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Standard of care + Radiation therapy (Experimental): Combination of N-803, ETBX-071, and M-CENK, along with radiation therapy.
  Interventions: Drug: N-803 (IL-15 Superagonist); Drug: ETBX-071 (PSA-based Oncolytic Virus); Drug: M-CENK (Activated NK Cells); Radiation: External Beam Radiation Therapy (EBRT); Radiation: Androgen Deprivation Therapy (ADT); Radiation: Post-radiation immunotherapy

INTERVENTIONS:
Drug: N-803 (IL-15 Superagonist) — Administered subcutaneously (SC) both before and after radiation therapy. The specific dosing schedule varies slightly depending on the cohort.
Drug: ETBX-071 (PSA-based Oncolytic Virus) — Administered subcutaneously (SC) before and after radiation therapy. The specific dosing schedule varies slightly depending on the cohort.
Drug: M-CENK (Activated NK Cells) — Administered intravenously (IV) before and after radiation therapy, also with variations in the timing and dosing across different cohorts.
Radiation: External Beam Radiation Therapy (EBRT) — This is a standard treatment administered to all participants. The specific dose and schedule (40 Gy in 5 fractions over 2 weeks or up to 9 weeks) are determined by the investigator based on clinical judgment.
Radiation: Androgen Deprivation Therapy (ADT) — May be used in conjunction with the other therapies. The specific type and duration of ADT are at the investigator's discretion, and it may be initiated up to 6 months after the completion of radiotherapy. This treatment is not part of the experimental treatment regimen.
Radiation: Post-radiation immunotherapy — The post-radiation immunotherapy phase in the ResQ110B-PROS study involves the continued administration of N-803, ETBX-071, and M-CENK, but with a specific schedule and after the completion of radiation therapy.

SUMMARY:
This study tests a new treatment for men with high-risk prostate cancer who can't have surgery. The treatment combines three experimental drugs and radiation therapy. Researchers will track how well the treatment works and how safe it is. The study will last about five years.

DETAILED DESCRIPTION:
This study (ResQ110B-PROS, IND 027158) is a Phase 2, open-label clinical trial designed to assess the safety and efficacy of a novel, multi-component treatment strategy for men with high-risk prostate cancer who are unsuitable for prostatectomy. The experimental treatment combines three investigational products with standard external beam radiation therapy (EBRT). The study is interventional, not observational.

The Investigational Products:

N-803 (nogapendekin alfa inbakicept): A soluble complex of an IL-15 variant bound to a human IL-15 receptor alpha subunit/human IgG1 Fc fusion protein. It acts as a growth and activation factor for NK cells and effector and memory T cells, aiming to stimulate the immune system's response to the cancer. Administered subcutaneously (SC).

ETBX-071 (hAd5 [E1-, E2b-, E3-]-PSA): A replication-defective human adenovirus serotype 5 (hAd5) vector modified to encode human prostate-specific antigen (PSA). This acts as a cancer vaccine, designed to generate an immune response targeting PSA-expressing prostate cancer cells. Administered subcutaneously (SC).

M-CENK (cytokine-induced memory-like NK cells): Autologous natural killer (NK) cells expanded and modified ex vivo using a cytokine cocktail (IL-12, IL-15, and IL-18) to enhance their cytotoxic activity and persistence. These cells are administered intravenously (IV).

Treatment Regimen:

The study employs a staged treatment approach:

Screening and Baseline Assessments: Participants undergo screening to confirm eligibility, including PSMA-PET scans, genomic testing, and PSA level assessment. Baseline assessments are collected before starting treatment.

Apheresis: Autologous peripheral blood mononuclear cells (MNCs) are collected from participants for the generation of M-CENK cells.

Pre-Radiation Immunotherapy: Participants receive N-803, ETBX-071, and M-CENK according to a specified schedule over a 6-week period. A targeted biopsy is performed before radiation.

Radiation Therapy (EBRT): Participants undergo EBRT (either a standard 2-week course or an extended 9-week course, as determined by the investigator).

Post-Radiation Immunotherapy: Following radiation, participants receive N-803, ETBX-071, and M-CENK for four 6-week cycles. Androgen deprivation therapy (ADT) may be initiated 6 months after completing radiotherapy.

Follow-up: Participants are followed for up to 5 years after the end of treatment (EOT).

Endpoints:

Primary: Complete pathologic response (CPR) after pre-radiation immunotherapy and PSA30 response at EOT after post-radiation immunotherapy.

Secondary: Clinical pathologic response, time to recurrence interval (TTRI), and safety.

Exploratory: Quality of life (QoL), sexual function, immune responses (including changes in immune subsets and antigen-specific responses), tumor microenvironment (TME), and circulating tumor DNA (ctDNA).

Study Population and Duration:

The study plans to enroll up to 20 participants. The total study duration is up to 303 weeks, including treatment and 5 years of follow-up.

ELIGIBILITY:
The inclusion criteria:

* Age: ≥18 years old.
* Ability to understand and provide informed consent: Participants must be able to understand the study and provide written informed consent fulfilling all relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
* Histologically confirmed prostate adenocarcinoma: A diagnosis confirmed through a pathology report or a clinical course consistent with the disease, as determined by a local pathologist, if a pathology specimen is unavailable.
* ECOG performance status: 0 or 1 (fully active or restricted in strenuous activity but ambulatory).
* Life expectancy: >5 years.
* Germline testing: Must have germline testing completed at the time of initial diagnosis and, if applicable, at recurrence.
* No evidence of distant metastasis: No evidence of soft tissue disease metastasis (visceral or lymph nodes) on CT/MRI scan.
* No active or organ-threatening autoimmune disease: Participants must not have an active or organ-threatening autoimmune disease.
* High-risk or very high-risk prostate cancer: Based on 2024 NCCN guidelines: PSA >20 ng/mL or Gleason Grade Group ≥4 or ≥cT3a.
* Adequate hematologic and organ function: Defined by specific laboratory values (ANC, lymphocyte count, platelet count, hemoglobin, INR/aPTT, AST, ALT, alkaline phosphatase) obtained within 14 days prior to baseline, with specific exceptions stated in the protocol for participants with liver or bone metastases or those with known Gilbert disease.
* Ability to attend study visits and return for adequate follow-up.
* Agreement to practice effective contraception: Non-sterile males must agree to use effective contraception (condom, vasectomy, or other barrier methods) for up to 7 months after treatment.

Exclusion Criteria:

* Prior treatment for prostate cancer: Participants who have undergone any prior surgical, cryotherapy, or high-intensity focused ultrasound treatment for prostate cancer are excluded.
* Prior hormonal therapy: Prior orchiectomy or hormonal therapy (GnRH agonists, NSAA) is an exclusion criterion.
* Prior treatment with androgen receptor (AR) inhibitors: Prior treatment with first-generation (bicalutamide, flutamide, nilutamide, cyproterone acetate) or second-generation (enzalutamide, apalutamide, or darolutamide) AR inhibitors is an exclusion criterion.
* Organ transplantation: Receipt of any organ transplantation (excluding those not requiring immunosuppression, such as corneal or hair transplants) excludes participants from the study.
* Chronic systemic corticosteroid use: Chronic administration (>14 days) of systemic corticosteroids within 28 days of study treatment initiation excludes participants. However, minimal systemic absorption (inhaled steroids, nasal sprays, topical agents) is permitted.
* Active autoimmune disease: Active autoimmune diseases (Addison's disease, Hashimoto's thyroiditis, systemic lupus erythematosus, Sjögren syndrome, scleroderma, myasthenia gravis, Goodpasture syndrome, or active Grave's disease) exclude participants. However, a history of autoimmunity that did not require systemic immunosuppression and did not threaten vital organ function is permitted.
* Use of medications affecting PSA: Use of medications known to alter PSA levels (5-alpha reductase inhibitors, phytoestrogens, saw palmetto) within 28 days before study treatment initiation excludes participants.
* Major surgery: Major surgery within 28 days of study treatment initiation excludes participants.
* Systemic therapy: Systemic therapy (including any investigational therapy) within 28 days of study treatment initiation is an exclusion criterion.
* Allergic reactions: A history of allergic reactions to compounds with similar chemical or biologic composition to the study drugs excludes participants.
* Clinically significant cardiovascular/cerebrovascular disease: This includes cerebral vascular accident/stroke, myocardial infarction, or unstable angina, congestive heart failure, or uncontrolled hypertension within specific timeframes before study enrollment.
* Serious intercurrent medical illness: Any serious intercurrent medical illness that could interfere with treatment participation.
* Active infections: Active HIV, hepatitis B (positive HBsAg), or hepatitis C infections exclude participation.
* Live attenuated vaccine administration: Administration of a live, attenuated vaccine within 3 weeks prior to study entry or anticipated during the study.
* Inability or unwillingness to comply: Participants assessed by the investigator as unable or unwilling to comply with the study requirements are excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete Pathologic Response (CPR) after pre-radiation immunotherapy. | CPR: Assessed within approximately 6 weeks of study start.
  Complete Pathologic Response (CPR) after pre-radiation immunotherapy: Assesses the complete absence of cancer in tissue samples taken after the pre-radiation immunotherapy phase. This signifies a complete eradication of the cancer at that stage of the treatment process.
PSA30 response at end-of-treatment (EOT) after post-radiation immunotherapy | Assessed at EOT, which occurs roughly 30 to 39 weeks after the study begins.
  Measures a ≥30% reduction in Prostate-Specific Antigen (PSA) levels from baseline to the end of treatment. PSA is a common biomarker used to monitor prostate cancer treatment success. A decrease in PSA suggests successful treatment in reducing the cancer burden.

SECONDARY OUTCOMES:
Clinical Pathologic Response (after pre-radiation immunotherapy) | Within approximately 6 weeks of the study start.
  Clinical Pathologic Response (CPR) is an assessment of the extent of tumor reduction after treatment, combining clinical (imaging) and pathological (tissue examination) findings. In this study, CPR is evaluated both after pre-radiation and post-radiation immunotherapy. The specific criteria for determining CPR will vary depending on whether it's assessed by imaging or pathology.
Time to Recurrence Interval (TTRI) | Variable, ranging from the end of radiation therapy (around 2-9 weeks after pre-radiation immunotherapy, depending on individual schedules) to up to 5 years (260 weeks).
  This measures the time elapsed between the completion of radiation therapy and the recurrence of the cancer. Longer TTRI indicates more durable treatment results.
Safety (AEs and SAEs) | Continuous monitoring throughout the entire study duration (approximately 303 weeks).
  Safety will be assessed by monitoring adverse events (AEs) and serious adverse events (SAEs) throughout the study, graded using the CTCAE v5.0 scale.

OTHER OUTCOMES:
Quality of Life (QoL) | Approximately 5 years
  Assessed using validated questionnaires
Sexual Function | Approximately 13 Months
  Assessed using the Sexual Health Inventory for Men (SHIM) questionnaire.
Changes in Immune Subsets and Antigen-Specific Immune Responses | Approximately 13 Months
  This evaluates the effects of the treatment on the immune system, looking for changes in various immune cells and their responses to specific cancer antigens.
PSA Levels | Approximately 13 months
  Prostate-specific antigen (PSA) is a protein produced by the prostate gland. PSA levels in the blood are commonly used as a marker to monitor prostate cancer.
Tumor Microenvironment (TME) | Pre-radiation TME: Approximately 6 weeks after study start. Post-radiation TME: Approximately 30-39 weeks after study start.
  Evaluated through analysis of tissue samples using whole slide images, spatial transcriptome, immunohistochemistry, and bulk RNA sequencing.
Circulating Tumor DNA (ctDNA) | Approximately 5 years
  Measured to assess the presence of cancer DNA in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, Study Chair — ImmunityBio, Inc.